CLINICAL TRIAL: NCT04952935
Title: Acupuncture for the Treatment of Medication-Dependent Hypotension in Heart Failure
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Scripps Health (Other)
Responsible Party: Principal Investigator, Yu-Ming Ni, Cardiology Fellow, Scripps Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-20-7569
Record Dates: First submitted 2021-05-21; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Congestive Heart Failure; Hypotension
Keywords: acupuncture; midodrine; fludrocortisone; randomized controlled trial
MeSH Terms: conditions — Heart Failure; Hypotension

STUDY DESIGN:
Intervention Model Description: Randomized double-blinded sham-controlled clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patient receives true or sham acupuncture, and patient is unaware of treatment assignment. Acupuncturist is aware of treatment assignment, as is the statistician who is aware of randomization assignment but not involved otherwise in the execution of clinical trial. Investigators, medical assistants, and patients' physicians are unaware of treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- True Acupuncture (Experimental)
  Interventions: Procedure: True Acupuncture
- Sham Acupuncture (Sham Comparator)
  Interventions: Procedure: Sham Acupuncture

INTERVENTIONS:
Procedure: True Acupuncture — Delivery of four acupuncture seeds (no needles involved) to the head and neck area at true acupuncture points.
  Arms: True Acupuncture
Procedure: Sham Acupuncture — Delivery of four acupuncture seeds (no needles involved) to the head and neck area at non-acupuncture points.
  Arms: Sham Acupuncture

SUMMARY:
Acupuncture is believed to increase blood pressure in people who struggle with low blood pressure. This is a common problem facing people with heart failure, and sometimes these people need to take medications to artificially increase their blood pressure. This study is designed to determine if using acupuncture in people with heart failure can improve their blood pressure enough to not require medications to artificially increase blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years old
* Chronic congestive heart failure (systolic or diastolic)
* Medication list includes midodrine or fludrocortisone, either taking as scheduled or as needed

Exclusion Criteria:

* History of acupuncture of any kind in the last 3 months
* Acute decompensated heart failure, as indicated by clinical picture at time of enrollment
* Currently on a mechanical device (LVAD, TAH, ECMO)
* History of hepatorenal syndrome, adrenal insufficiency, for which midodrine and fludrocortisone respectively is specifically being used to treat that condition
* Lack of suitable locations for which to place acupuncture seeds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | 9 weeks
  Change in mean arterial blood pressure, as measured by blood pressure cuff in sitting position

SECONDARY OUTCOMES:
Blood Pressure adjusted for Medication | 9 weeks
  Change in mean arterial blood pressure, as measured by blood pressure cuff in sitting position, adjusted for midodrine/fludrocortisone dose as covariate
Standing Blood Pressure adjusted for Medication | 9 weeks
  Change in mean arterial blood pressure, as measured by blood pressure cuff in standing position, adjusted for midodrine/fludrocortisone dose as covariate
Medication Dose Change | 9 weeks
  Percentage change in median dose of midodrine or fludrocortisone (in mg per week)
Got off medications | 9 weeks
  Number of patients who came off of midodrine or fludrocortisone by end of study
NYHA Class | Start, 5 weeks, and 9 weeks
  Change in NYHA Class
Quality of Life Score | Start, 5 weeks, and 9 weeks
  Change in Quality of Life scores by VAS
Composite Safety Outcome | Throughout study, total time 9 weeks
  Composite of skin injury, symptomatic hypotension, hospitalization for heart failure exacerbation or syncope or hypotension, implantation of LVAD/MCS device or heart transplantation, or all-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Suhar, MD, Principal Investigator — Scripps Health; Yu-Ming Ni, MD, Principal Investigator — Scripps Health; Rajeev Mohan, MD, Principal Investigator — Scripps Health
Locations (2):
- United States (2):
  - Scripps La Jolla Medical Center, La Jolla, California
  - Scripps Shiley Integrative Center, La Jolla, California